CLINICAL TRIAL: NCT00130598
Title: PROVOCATION Trial - PROphylactic intraVenOus Hydration for Contrast Agent Toxicity PreventION
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: University Hospital, Basel, Switzerland, Christian Mueller, MD
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PROVOCATION Trial; 23.05; 05.013; 2005DR3170
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Last update posted 2010-03-05 (Estimated); Status verified 2010-03

CONDITIONS: Kidney Failure, Acute
Keywords: contrast nephropathy; contrast media; renal dysfunction
MeSH Terms: conditions — Acute Kidney Injury; Renal Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): control group: patients receive a preventive hydration with 154mEq/l saline at an ongoing rate of 1ml/kg per hour of at least 12 hours prior and after the procedure.
  Interventions: Drug: NaCl 0.9% i.v. or NaBic 1.4% i.v. or NaBic 1.4% i.v. + NaBic p.o. (Nephrotrans®)
- 2 (Active Comparator): 7h-sodium bicarbonate (according to the regimen used in a recently published study (slightly modified)14): before contrast a bolus of 3ml/kg NaHCO3 166mEq/l for one hour, followed by an infusion of NaHCO3 166mEq/l with a rate of 1ml/kg per hour until 6h after contrast.
  Interventions: Drug: NaCl 0.9% i.v. or NaBic 1.4% i.v. or NaBic 1.4% i.v. + NaBic p.o. (Nephrotrans®)
- 3 (Active Comparator): short-term sodium bicarbonate: NaHCO3 166mEq/l (3ml/kg; patients with a body weight above 100kg 300ml) as a bolus 20 minutes before contrast; additionally ingestion of Nephrotrans® (500mg NaHCO3/capsule: 1 capsule/10kg) with 1-2 dl of San Pellegrino® non-sparkling mineral water at the start of the infusion. Ingestion of 500ml San Pellegrino® non-sparkling mineral water in the first 6 hours after contrast.
  Interventions: Drug: NaCl 0.9% i.v. or NaBic 1.4% i.v. or NaBic 1.4% i.v. + NaBic p.o. (Nephrotrans®)

INTERVENTIONS:
Drug: NaCl 0.9% i.v. or NaBic 1.4% i.v. or NaBic 1.4% i.v. + NaBic p.o. (Nephrotrans®) — control group: preventive hydration with 154mEq/l saline at 1ml/kg per hour of 12 hours prior and after the procedure.
  7h-sodium bicarbonate: before contrast 3ml/kg NaHCO3 166mEq/l for one hour, followed by NaHCO3 166mEq/l (1ml/kg per hour until 6h after contrast).
  short-term sodium bicarbonate: NaHCO3 166mEq/l (3ml/kg) as a bolus 20 minutes before contrast; ingestion of Nephrotrans® (500mg NaHCO3/capsule: 1 capsule/10kg) with 1-2 dl non-sparkling mineral water at the start of the infusion. Ingestion of non-sparkling mineral water in the first 6 hours after contrast.
  Other Names: NaCl 0.9% Braun®; NaBic 1.4% Bichsel®; Nephrotrans®

SUMMARY:
Contrast nephropathy (CN) remains a common complication of radiographic procedures and an important cause of hospital-acquired acute renal failure. Only hydration with saline is uniformly accepted and used in clinical practice as a cornerstone for the prevention of CN. But the optimal preventive strategy for CN is not known. Sodium bicarbonate might be even more effective than hydration with sodium chloride for prophylaxis of CN. Therefore the aim of the study is to evaluate the efficacy of two regimens of sodium bicarbonate compared with a prolonged infusion of sodium chloride in the prevention of CN.

Primary endpoint: Decrease in glomerular filtration rate (GFR) within 48 hours.

DETAILED DESCRIPTION:
Background: Contrast nephropathy (CN) remains a common complication of radiographic procedures and an important cause of hospital-acquired acute renal failure, which contributes to morbidity and mortality during hospitalization, as well as costs of health care. Many previous strategies to prevent CN (such as N-acetylcysteine, aminophylline, fenoldopam, hemofiltration) have been unsuccessful or at least controversial. Only hydration with saline is uniformly accepted and used in clinical practice as cornerstone for the prevention of CN. But the optimal preventive strategy for CN is not known. According to a recent study, periprocedural hydration with sodium bicarbonate might be even more effective than hydration with sodium chloride for prophylaxis of CN. Such a preventive hydration with sodium bicarbonate should be compared with the gold standard of hydration with saline (24-h hydration period). This has not been evaluated so far. Given its high oral bioavailability, sodium bicarbonate could be administered even orally instead of a prolonged infusion. An effective short-term regimen would be highly attractive in clinical practice including outpatient procedures.

Aim: To evaluate the efficacy of two regimens of sodium bicarbonate compared with a prolonged infusion of sodium chloride in the prevention of CN.

Primary endpoint: Decrease in glomerular filtration rate (GFR) within 48 hours. GFR is calculated using the abbreviated Modification of Diet in Renal Disease Study equation. Secondary endpoints: Development of contrast nephropathy defined by increase in serum creatinine concentration of at least 44umol/l within 48 hours, an increase >=25% in the baseline serum creatinine concentration within 48 hours, or defined as an increase >=25% in the baseline serum cystatin C concentration or an increase >=0.35mg/l in serum cystatin C concentration within 48 hours; increase in serum cystatin C level at day 1 and 2, in-hospital morbidity (nonfatal myocardial infarction) and mortality, dialysis, length of stay, total costs of hospitalization, 3-/12-month mortality, 3-/12-month hospitalization for cardiac causes, and GFR at 3 and 12 months.

Patients and Methods: This randomized, controlled open-label trial is designed to enroll 258 patients at increased risk for CN because of renal dysfunction undergoing intraarterial or intravenous radiographic contrast procedures. Patients will be randomly assigned 1:1:1 with the use of sealed envelopes into 3 groups (block randomisation for intraarterial and intravenous radiographic contrast procedures) :

1. a control group: patients receive a preventive hydration with 154mEq/l saline at an ongoing rate of 1ml/kg per hour of at least 12 hours prior and after the procedure.
2. a group with 7h-sodium bicarbonate (according to the regimen used in a recently published study (slightly modified)14): before contrast a bolus of 3ml/kg NaHCO3 166mEq/l for one hour, followed by an infusion of NaHCO3 166mEq/l with a rate of 1ml/kg per hour until 6h after contrast.
3. a group with short-term sodium bicarbonate: NaHCO3 166mEq/l (3ml/kg; patients with a body weight above 100kg 300ml) as a bolus 20 minutes before contrast; additionally ingestion of Nephrotrans® (500mg NaHCO3/capsule: 1 capsule/10kg) with 1-2 dl of San Pellegrino® non-sparkling mineral water at the start of the infusion. Ingestion of 500ml San Pellegrino® non-sparkling mineral water in the first 6 hours after contrast.

Expected results: It is the researchers' hypothesis that a short-term periprocedural preventive hydration with sodium bicarbonate will be non-inferior to the regimen of long-term hydration with sodium bicarbonate. The long-term regimen with sodium bicarbonate is expected to be superior to the standard i.v. regimen with sodium chloride.

Significance: Given the significant morbidity and mortality associated with acute renal failure due to contrast media as well as the widespread use of contrast media in an ambulant setting for diagnostic and therapeutical procedures, preventive short-term hydration with sodium bicarbonate could represent a major advance in clinical medicine.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted with renal dysfunction (baseline serum creatinine level above the upper limit of normal of the serum creatinine [>93umol/l for women and >117umol/l for men] or GFR <60ml/min [GFR calculated using the abbreviated MDRD study equation]) scheduled to undergo an intraarterial or intravenous radiographic contrast procedure within the next 24 hours.

Exclusion Criteria:

* Age <18 years
* Preexisting dialysis
* Allergy to radiographic contrast
* Pregnancy (women < 50 years: pregnancy test required)
* Severe heart failure (New York Heart Association [NYHA] III-IV)
* N-acetylcysteine </= 24 hours before contrast
* Clinically vulnerable condition requiring continuous fluid therapy e.g. severe sepsis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Actual)
Dates: Start 2005-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Decrease in glomerular filtration rate (GFR) within 48 hours. GFR is calculated using the abbreviated Modification of Diet in Renal Disease (MDRD) Study equation. | 48 hours

SECONDARY OUTCOMES:
Development of contrast nephropathy, defined as an increase >=25% in the baseline serum creatinine concentration within 48 hours | 48 hours
Development of contrast nephropathy, defined as an increase >=44umol/l in serum creatinine concentration within 48 hours | 48 hours
Development of contrast nephropathy, defined as an increase >=25% in the baseline serum cystatin C concentration or an increase >=0.35mg/l in serum cystatin C concentration within 48 hours | 48 hours
Postcontrast increase in serum cystatin C at day 1 and 2 | 48 hours
In-hospital morbidity (nonfatal myocardial infarction) and mortality | 60 days
Dialysis dependency | 12 months
Length of stay | 60 days
Total costs of hospitalization | 60 days
3-/12-month mortality | 12 months
3-/12-month hospitalization for cardiac causes | 12 months
GFR at 3 and 12 months | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Christian Mueller, Prof., Principal Investigator — University Hospital of Basel
Locations (3):
- Centro Cardiologico Monzino, Milan, Italy
- Switzerland (2):
  - University Hospital of Basel, Basel, Basel
  - Kantonsspital Liestal - Universitätskliniken, Liestal

REFERENCES:
- [Background] Merten GJ, Burgess WP, Gray LV, Holleman JH, Roush TS, Kowalchuk GJ, Bersin RM, Van Moore A, Simonton CA 3rd, Rittase RA, Norton HJ, Kennedy TP. Prevention of contrast-induced nephropathy with sodium bicarbonate: a randomized controlled trial. JAMA. 2004 May 19;291(19):2328-34. doi: 10.1001/jama.291.19.2328. PMID 15150204
- [Background] Mueller C, Seidensticker P, Buettner HJ, Perruchoud AP, Staub D, Christ A, Buerkle G. Incidence of contrast nephropathy in patients receiving comprehensive intravenous and oral hydration. Swiss Med Wkly. 2005 May 14;135(19-20):286-90. doi: 10.4414/smw.2005.10938. PMID 15986266
- [Background] Mueller C, Buerkle G, Buettner HJ, Petersen J, Perruchoud AP, Eriksson U, Marsch S, Roskamm H. Prevention of contrast media-associated nephropathy: randomized comparison of 2 hydration regimens in 1620 patients undergoing coronary angioplasty. Arch Intern Med. 2002 Feb 11;162(3):329-36. doi: 10.1001/archinte.162.3.329. PMID 11822926
- [Derived] Klima T, Christ A, Marana I, Kalbermatter S, Uthoff H, Burri E, Hartwiger S, Schindler C, Breidthardt T, Marenzi G, Mueller C. Sodium chloride vs. sodium bicarbonate for the prevention of contrast medium-induced nephropathy: a randomized controlled trial. Eur Heart J. 2012 Aug;33(16):2071-9. doi: 10.1093/eurheartj/ehr501. Epub 2012 Jan 19. PMID 22267245
- See also: Related Info — http://www.dyspnea.ch